CLINICAL TRIAL: NCT04889560
Title: Home-based Cognitive Treatment of Early Stages of Cognitive Impairment in Neurodegenerative Diseases: Home CoRe
Brief Title: Home-based Cognitive Treatment and Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Home CoRe 2021
Record Dates: First submitted 2021-05-07; First posted 2021-05-17 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2021-05

CONDITIONS: Cognitive Impairment
Keywords: Neurodegenerative disease; Cognitive decline; Non-pharmacological treatments; Cognitive training; Home-based CT
MeSH Terms: conditions — Cognitive Dysfunction; Neurodegenerative Diseases | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (neuropsychologist for cognitive assessments)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group receives Home CoRe (Home CoRe Group)
  Interventions: Other: Experimental group
- Control group (Other): Control group receives CoRe software (CoRe Group)
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental group — Home-based version of a computerized cognitive training (CoRe)
  Arms: Experimental group
Other: Control group — Computerized cognitive training (CoRe)
  Arms: Control group

SUMMARY:
The prevalence of neurodegenerative diseases is expected to increase over the next years, in parallel with the aging of the world population. Therefore, it is important to identify new methods to prevent, delay or stop the neurodegenerative waterfall responsible for dementia conversion. To date, there is no fully proven pharmacological treatment for cognitive impairment and the available pharmacological treatments have limited efficacy because consist in symptomatic drugs with adverse side effects. On this point, non-pharmacological intervention may represent adjunctive therapy to medications in order to prevent or delay the onset of the cognitive deficits or dementia. Recently we evaluated the effectiveness of a computerized cognitive training (CoRe) in patients with early cognitive impairment. The main goal of the present protocol is to evaluate the efficacy of the home-based version of CoRe (Home CoRe). To this end, mild dementia or early cognitive impairment, and persons with Subjective Cognitive Impairment (SCI) are enrolled and randomly assigned to the experimental group (Home CoRe) or control group (CoRe). All patients are evaluated before (T0) and after (T1) treatment with an exhaustive neuropsychological assessment. Furthermore, follow-up visits are scheduled 6 months (T2) and 12 months (T3) after the end of the treatment.

DETAILED DESCRIPTION:
Non-pharmacological intervention may represent adjunctive therapy to medications in order to delay the onset of the cognitive deficits or dementia. Moreover, increasing evidence suggests that environmental and lifestyle factors (education, cognitive engagement, experience..) impact on cognitive functions and brain plasticity during the lifetime and also during aging. These modifiable factors moderate differences in cognitive aging and are protective for the development of dementia.

Among non-pharmacological approaches, previous studies observed a positive effect of Cognitive Training (CT) both in healthy elderly people and patients in the early stage of neurodegenerative diseases. Moreover, the advances in the development of Information & Communication Technologies (ICT) has prompted the possibility to develop computer-based solution for the training of cognitive functions, being able to overcome traditional-training advantages. However, some issue remain unresolved and larger randomized controlled trials are necessary to examine long-term CT effects, due to the lack of longitudinal studies. Our previous data demonstrated that CT program with CoRe software is safe and effective on cognition in patient with Parkinson Disease-Mild Cognitive Impairment, in the attempt of briefly stabilizing cognitive decline, delaying the downward trajectory. The same pattern of findings resulted when using CoRe in patients with Mild Cognitive Impairment (MCI) and mild Alzheimer's Disease (AD). Among ICT advantages there is the fact that they offer the possibility to develop patient tailored interventions that can be easily delivered not only in-person but also remotely at patients' homes. It means that they could simplify the therapist's work in terms of the planning, design, and management of the cognitive intervention also outside from the clinical setting. However, some concerns have slowed the integration of home-based interventions into clinical practice, such as the fact that people with advanced age or cognitive deficit might have poor computer skills and difficulties managing technological devices on their own. Thus, the overall efficacy of home-based CT programs is still under debate.

In this frame, the primary goal of this single-blind randomized controlled trial is to assess whether a home-based CT (Home CoRe) could offer comparable effects (non-inferiority trial) to those of an in-person CT (CoRe). A secondary goal is to follow these effects with respect to the evolution of cognitive decline. These two interventions are evaluated also in terms of treatment adherence.

Both treatment protocols consist of 18 sessions (3 session/week, 45 minutes/day) of CT with CoRe vs HomeCoRe software (training memory and logical-executive functions).

Patients with mild dementia, early cognitive impairment (i.e., MCI and vascular cognitive impairment (VCI)), and SCI are recruited from Neuropsychology/Alzheimer's Disease Assessment Unit and Neurorehabilitation Unit of IRCCS Mondino Foundation. Patients' diagnosis is formulated on the basis of a comprehensive neuropsychological evaluation (baseline cognitive assessment - T0) according to the guidelines presented in the literature. The following standardized tests assessing different domains are used:

* global cognitive function: Mini-Mental State Examination (MMSE) and Montreal Montreal Overall Cognitive Assessment (MoCA);
* memory: verbal (Verbal Span; Digit Span) and spatial (Corsi's blocktapping test - CBTT) span; verbal long-term memory (Logical Memory Test immediate and delayed recall; Rey's 15-word test immediate and delayed recall); spatial long-term memory (Rey Complex Figure delayed recall - RCF-dr);
* logical-executive functions: non-verbal reasoning (Raven's Matrices 1947 - RM47); frontal functionality (Frontal Assessment Battery - FAB); semantic fluency (animals, fruits, car brands), phonological fluency (FAS);
* attention: visual selective attention (Attentive Matrices); simple speed processing and complex attention (Trail Making Test parts A - TMT A and part B - TMT B);
* visuospatial abilities: constructive apraxia Rey Complex Figure copy - RCF-copy.

The same battery is also used at follow-up visits; parallel versions are applied when available (verbal long-term memory tests), in order to avoid the learning effect. All the test scores are corrected for age, sex, and education and compared with the values available for the Italian population.

At the baseline, the cognitive reserve is assessed using Cognitive Reserve Index questionnaire (CRIq). The patients' functional status is assessed using Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) at the baseline and at the last follow-up visit after one year (T3). Moreover, mood is assessed using the Beck Depression Inventory (BDI) at the baseline and at the follow-up visits (T1, T2 and T3), while quality of life were assessed using the 36-Item Short Form Health Survey questionnaire (SF-36) at the baseline and at the follow-up visits six months (T2) and one year (T3) after training. Subjective evaluation of intervention success is also considered by means of the Patient Global Impression of Change (PGIC) and the Patients Reported Outcome Measures (PROMS), administered at T0 and T1. Treatment adherence is evaluated considering the number of CT sessions carried out.

All the patients recruited undergo baseline cognitive assessment (T0). Patients who met the inclusion and exclusion criteria are enrolled and randomly assigned to the experimental group (Home CoRe) or control group (CoRe).

ELIGIBILITY:
Inclusion Criteria:

* presence of mild dementia, mild cognitive impairment; vascular cognitive impairment, subjective cognitive impairment;
* age between 50 and 85 years;
* educational level ≥ 5 years.

Exclusion Criteria:

* MMSE < 20
* CRD > 1
* pre-existing cognitive impairment (e.g. aphasia, neglect);
* severe disturbances in consciousness;
* concomitant severe psychiatric disease or others neurological conditions (e.g. depression and behavioral disorders).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Change from T0 to T1, T2 and T3
  Global cognitive functioning measured by MMSE. MMSE is a neuropsychological test for the evaluation of intellectual efficiency disorders and the presence of cognitive impairment. The total score is between a minimum of 0 and a maximum of 30 points. A score of 18 or less indicates a severe impairment of cognitive abilities a score between 18 and 24 indicates moderate to mild impairment, a score of 25 is considered borderline, and a score of 26 to 30 indicates cognitive normality.
Montreal Overall Cognitive Assessment (MoCA) | Change from T0 to T1, T2 and T3
  Global cognitive functioning measured by MoCA. MoCA is a widely used screening assessment for detecting cognitive impairment. The MoCA test is a 30-point test. Lower score is worst outcome.

SECONDARY OUTCOMES:
Beck Depression Inventory - BDI | Change from T0 to T1, T2 and T3
  Mood assessed by BDI. BDI is a 21-question multiple-choice self-report inventory. Higher total scores indicate more severe depressive symptoms. Each question has a set of at least four possible responses, ranging in intensity. Higher total scores indicate more severe depressive symptoms.
Short Form-36 Health Survey - SF-36 | Change from T0 to T1, T2 and T3
  Quality of life assessed by SF-36. The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health.
Patient Global Impression of Change - PGIC | Change from T0 to T1
  Subjective evaluation of intervention success assessed by PGIC. The self-report measure PGIC reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement.
Patients Reported Outcome Measures (PROMS) | Change from T0 to T1
  Subjective evaluation of intervention success assessed by PROMS. PROMs are used to assess a patient's health status at a particular point in time. PROMs tools can be completed either during an illness or while treating a health condition. In some cases, using pre- and post-event PROMs can help measure the impact of an intervention.
Number of CT sessions completed | Change from T0 to T1, T2 and T3
  Treatment adherence assessed by number of cognitive training sessions completed.
Clinical Dementia Rating Scale (CDR) | Change from T0 to T1, T2 and T3
  The evolution of cognitive profile assessed by CDR. The CDR Dementia Staging Instrument in one aspect is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Cappa, Prof, Principal Investigator — IRCCS Mondino Foundation, Pavia
Locations (1):
- Dementia Research Center, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Coyle H, Traynor V, Solowij N. Computerized and virtual reality cognitive training for individuals at high risk of cognitive decline: systematic review of the literature. Am J Geriatr Psychiatry. 2015 Apr;23(4):335-359. doi: 10.1016/j.jagp.2014.04.009. Epub 2014 May 14. PMID 24998488
- [Background] Hachinski V, Iadecola C, Petersen RC, Breteler MM, Nyenhuis DL, Black SE, Powers WJ, DeCarli C, Merino JG, Kalaria RN, Vinters HV, Holtzman DM, Rosenberg GA, Wallin A, Dichgans M, Marler JR, Leblanc GG. National Institute of Neurological Disorders and Stroke-Canadian Stroke Network vascular cognitive impairment harmonization standards. Stroke. 2006 Sep;37(9):2220-41. doi: 10.1161/01.STR.0000237236.88823.47. Epub 2006 Aug 17. PMID 16917086
- [Background] Hsu WY, Ku Y, Zanto TP, Gazzaley A. Effects of noninvasive brain stimulation on cognitive function in healthy aging and Alzheimer's disease: a systematic review and meta-analysis. Neurobiol Aging. 2015 Aug;36(8):2348-59. doi: 10.1016/j.neurobiolaging.2015.04.016. Epub 2015 May 1. PMID 26022770
- [Background] Lampit A, Hallock H, Valenzuela M. Computerized cognitive training in cognitively healthy older adults: a systematic review and meta-analysis of effect modifiers. PLoS Med. 2014 Nov 18;11(11):e1001756. doi: 10.1371/journal.pmed.1001756. eCollection 2014 Nov. PMID 25405755
- [Background] Livingston G, Sommerlad A, Orgeta V, Costafreda SG, Huntley J, Ames D, Ballard C, Banerjee S, Burns A, Cohen-Mansfield J, Cooper C, Fox N, Gitlin LN, Howard R, Kales HC, Larson EB, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care. Lancet. 2017 Dec 16;390(10113):2673-2734. doi: 10.1016/S0140-6736(17)31363-6. Epub 2017 Jul 20. No abstract available. PMID 28735855
- [Background] Mendonca MD, Alves L, Bugalho P. From Subjective Cognitive Complaints to Dementia: Who is at Risk?: A Systematic Review. Am J Alzheimers Dis Other Demen. 2016 Mar;31(2):105-14. doi: 10.1177/1533317515592331. PMID 26142292
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Prehn K, Floel A. Potentials and limits to enhance cognitive functions in healthy and pathological aging by tDCS. Front Cell Neurosci. 2015 Sep 14;9:355. doi: 10.3389/fncel.2015.00355. eCollection 2015. PMID 26441526
- [Background] Sachdev PS, Blacker D, Blazer DG, Ganguli M, Jeste DV, Paulsen JS, Petersen RC. Classifying neurocognitive disorders: the DSM-5 approach. Nat Rev Neurol. 2014 Nov;10(11):634-42. doi: 10.1038/nrneurol.2014.181. Epub 2014 Sep 30. PMID 25266297
- [Result] Bernini S, Alloni A, Panzarasa S, Picascia M, Quaglini S, Tassorelli C, Sinforiani E. A computer-based cognitive training in Mild Cognitive Impairment in Parkinson's Disease. NeuroRehabilitation. 2019;44(4):555-567. doi: 10.3233/NRE-192714. PMID 31256092
- [Result] Bernini S, Panzarasa S, Barbieri M, Sinforiani E, Quaglini S, Tassorelli C, Bottiroli S. A double-blind randomized controlled trial of the efficacy of cognitive training delivered using two different methods in mild cognitive impairment in Parkinson's disease: preliminary report of benefits associated with the use of a computerized tool. Aging Clin Exp Res. 2021 Jun;33(6):1567-1575. doi: 10.1007/s40520-020-01665-2. Epub 2020 Sep 8. PMID 32895890
- [Derived] Bernini S, Valcarenghi A, Panzarasa S, Quaglini S, Costa A, Ramusino MC, Picascia M, Barbieri M, Tassorelli C, Vecchi T, Bottiroli S. HomeCoRe for telerehabilitation in mild or major neurocognitive disorders: a non-inferiority randomized controlled trial. Geroscience. 2025 Nov 13. doi: 10.1007/s11357-025-02006-9. Online ahead of print. PMID 41225283
- [Derived] Bernini S, Panzarasa S, Sinforiani E, Quaglini S, Cappa SF, Cerami C, Tassorelli C, Vecchi T, Bottiroli S. HomeCoRe for Telerehabilitation in Mild or Major Neurocognitive Disorders: A Study Protocol for a Randomized Controlled Trial. Front Neurol. 2021 Dec 23;12:752830. doi: 10.3389/fneur.2021.752830. eCollection 2021. PMID 35002919